CLINICAL TRIAL: NCT00385918
Title: Cardiovascular Parameters for Lokomat Training in Chronic Incomplete SCI
Brief Title: Robotically Assisted Treadmill Training in Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Maryland (Other); Kernan Orthopaedics and Rehabilitation Hospital (Unknown)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B4027; B40271 (Other: UMB-IRB old BRAAN system); HP-00042597 (Other: UMB-IRB)
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-04

CONDITIONS: Paraplegia; Quadriplegia; Spinal Cord Injury; Tetraplegia
Keywords: Cardiovascular Fitness; Exercise; Gait; Spinal Cord Injury; Treadmill Training
MeSH Terms: conditions — Paraplegia; Quadriplegia; Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lokomat training (Experimental): Subjects will receive active exercise treatment in the Lokomat device 3 times per week for 3 months. Each session will last approximately 45 minutes.
  Interventions: Device: Lokomat Training
- Home stretching then Lokomat training (Active Comparator): Patients will participate in a home stretching program for 3 months. They will then be crossed over to an active Lokomat treatment for a subsequent 3 months.
  Interventions: Other: Home stretching then Lokomat training

INTERVENTIONS:
Device: Lokomat Training — The Lokomat is a robotically assisted partial weight suspension treadmill training device that has the potential to restore leg function in persons with incomplete leg paralysis.
  Arms: Lokomat training
Other: Home stretching then Lokomat training — Patients will be instructed by a physical therapist on how to perform a home stretching protocol 3 times per week for 3 months. The stretching will be monitored via telephone by the study coordinator. This will be an active control arm. After 3 months the patients will be crossed over to Lokomat training for an additional 3 months. This training will be the same as given to the individuals originally randomized to the Lokomat treatment intervention.
  Arms: Home stretching then Lokomat training

SUMMARY:
This proposal investigates the hypothesis that progressive aerobic exercise with Lokomat is feasible in people with motor incomplete spinal cord injury, and three months of training will improve cardiovascular fitness and gait functionality when compared to physical therapy controls

DETAILED DESCRIPTION:
Little information is available about the cardiovascular effects of robotically assisted partial weight support treadmill training devices such as Lokomat in chronic incomplete spinal cord injured subjects. Task-oriented aerobic exercise has the potential to improve both neuromuscular function and cardiovascular metabolic fitness in neurological populations. Since spinal cord injured individuals are at an increased risk of developing premature cardiovascular disease, the investigation of robotic-assisted interventions in spinal cord injury (SCI) such as the Lokomat may have important health benefits in both cardiovascular fitness as well as functional mobility.

This proposal investigates the hypothesis that progressive aerobic exercise with Lokomat is feasible in motor incomplete SCI, and three months of training will improve cardiovascular fitness and gait functionality when compared to physical therapy controls. We propose a two-phase study to examine the feasibility, reliability and utility of aerobic exercise metabolic testing and training during robotically assisted partial weight support treadmill walking in individuals with chronic motor incomplete spinal cord injury (CMISCI). During the first phase of the study we will manipulate Lokomat training parameters of treadmill speed and percent of partial weight support to assess the effect of these changes on heart rate, perceived exertion, and oxygen consumption in untrained chronic motor incomplete spinal cord injured subjects. Subjects will be asked to maintain cardiovascular or muscular effort during testing and will be monitored in this regard by the force biofeedback system built into the Lokomat. After determining threshold levels for initial cardiovascular response, submaximal and then peak exercise testing will be attempted. These studies will be repeated on a separate day to determine the reliability of the testing results. Thirty-six subjects with varying levels of injury between C4 and L2 and ASIA (American Spinal Injury) Impairment Scales of C and D will be recruited. We anticipate that subjects with greater ASIA motor scores will require either a faster initial treadmill speed or less partial weight support to produce an initial cardiovascular response. It is also anticipated that peak exercise testing using open circuit spirometry with subjects on the Lokomat will be a feasible, reliable and valid measurement. This phase of the study will be aimed at establishing guidelines for determining initial training parameters for use in an aerobic exercise protocol using the Lokomat.

The second phase of this pilot study will be a controlled trial of three-month progressive aerobic Lokomat exercise in chronic incomplete spinal cord injured subjects. The aim of this trial will be to determine whether progressive Lokomat training will improve cardiovascular fitness and ambulatory function when compared to matched impairment severity CMISCI subjects receiving the same duration of usual physical therapy care. Thirty-six subjects will be recruited into this phase of the study. Open spirometric evaluation of cardiovascular parameters as outlined in phase one of the proposal will be measured at baseline, 1 months, and 3 months. Initial, six-week and post-study ambulatory function evaluations including the WISCI (Walking Index for Spinal Cord Injury), a timed 10 meter walk, a measured walk over 6 minutes, and a gait analysis will also be determined. It is hypothesized that aerobic Lokomat exercise will improve cardiovascular fitness as determined by an increase in VO2 (oxygen consumption) peak and improve function as determined by timed walks and gait parameters in these subjects. The results of this pilot and development study will provide the necessary information to design larger randomized clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset Spinal Cord Injury or Disease at least 12 months prior to enrollment
* Age 18 to 80
* Level of injury from C4 to L2
* ASIA impairment scale either C or D
* Able to tolerate standing frame for at least 30 minutes

Exclusion Criteria:

* History of unstable angina, recent MI (myocardial infarction), CHF (congestive heart failure) or clinically significant valvular dysfunction
* History of recent hospitalization (<3 months) for a major medical problem

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gorman, MD MS, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (2):
- United States (2):
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - University of Maryland Rehabilitation and Orthopaedic Institute, Baltimore, Maryland

REFERENCES:
- [Result] Gorman PH, Geigle PR, Chen K, York H, Scott W. Reliability and relatedness of peak VO2 assessments during body weight supported treadmill training and arm cycle ergometry in individuals with chronic motor incomplete spinal cord injury. Spinal Cord. 2014 Apr;52(4):287-91. doi: 10.1038/sc.2014.6. Epub 2014 Feb 18. PMID 24534779
- [Derived] Gorman PH, Scott W, York H, Theyagaraj M, Price-Miller N, McQuaid J, Eyvazzadeh M, Ivey FM, Macko RF. Robotically assisted treadmill exercise training for improving peak fitness in chronic motor incomplete spinal cord injury: A randomized controlled trial. J Spinal Cord Med. 2016;39(1):32-44. doi: 10.1179/2045772314Y.0000000281. Epub 2014 Dec 18. PMID 25520035
- See also: Website of the manufacturer of the Lokomat — http://www.hocoma.com
- See also: Hospital where the research is being undertaken. — http://www.kernan.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: April 2007 through 2010. Location of recruitment: Kernan Hospital Spinal Cord Injury Clinic and Baltimore VAMC Spinal Cord Support Clinic.
Pre-assignment Details: Participants all underwent baseline and feasibility testing prior to randomization in either of the two arms.
Groups:
- Lokomat Training: Subjects will receive active exercise treatment in the Lokomat device 3 times per week for 3 months. Each session will last approximately 45 minutes.
  Lokomat Training : The Lokomat is a robotically assisted partial weight suspension treadmill training device that has the potential to restore leg function in persons with incomplete leg paralysis.
- Home Stretching Then Lokomat Training: Patients will participate in a home stretching program for 3 months.
  Home stretching protocol : Patients will be instructed by a physical therapist on how to perform a home stretching protocol 3 times per week for 3 months. The stretching will be monitored via telephone by the study coordinator. This will be an active control arm.
  After 3 months the participants will be switched to a 3 month period of Lokomat training the same as that offered to the patients randomized to the "Lokomat Training" arm of the study.
- Baseline and Feasibility Testing: All subjects were screened and underwent baseline testing prior to randomization into either the Lokomat training or the Home stretching then Lokomat training group.
Period: Feasibility & Baseline Measurement Phase
Arm/Group | Lokomat Training | Home Stretching Then Lokomat Training | Baseline and Feasibility Testing
Started | 0 | 0 | 35 (Total # of subjects screened.The screening occurred before randomization.)
Number Eligible | 0 | 0 | 27 (8 subjects failed screening.)
Completed Baseline Tests | 0 | 0 | 21 (6 subjects did not complete all baseline tests.)
Completed | 0 | 0 | 21
Not Completed | 0 | 0 | 14
Not completed — outside of inclusion criteria | 0 | 0 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 5
Not completed — Physician Decision | 0 | 0 | 1
Period: Intervention Phase After Randomization
Arm/Group | Lokomat Training | Home Stretching Then Lokomat Training | Baseline and Feasibility Testing
Started | 15 (Participant successfully completed screening; this is the number in the Lokomat training arm.) | 6 (Participants successfully completed screening; this is the number in the home stretching arm.) | 0
Completed | 12 (Participants completed the 3-month training intervention) | 6 (Participants completed the 3-month home-base intervention) | 0
Not Completed | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis includes data from individuals who have completed the 3-month robotic and home-base interventions
Groups:
- Lokomat Exercise: Subjects will receive active exercise treatment in the Lokomat device 3 times per week for 3 months. Each session will last approximately 45 minutes.
  Lokomat Training : The Lokomat is a robotically assisted partial weight suspension treadmill training device that has the potential to restore leg function in persons with incomplete leg paralysis.
- Home Stretching Then Lokomat Exercise: Patients will participate in a home stretching program for 3 months. They will then be crossed over to Lokomat treatment for an additional 3 months.
  Home stretching protocol : Patients will be instructed by a physical therapist on how to perform a home stretching protocol 3 times per week for 3 months. The stretching will be monitored via telephone by the study coordinator. This will be an active control arm.
- Total: Total of all reporting groups
Arm/Group | Lokomat Exercise | Home Stretching Then Lokomat Exercise | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.7) | 52.0 (15.4) | 51.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 11 | 6 | 17
Lower Extremity Motor Score [Mean (Standard Deviation); unit: units on a scale] — The motor score assigned to the five key bi-lateral lower extremity muscle groups with values ranging from 0 (total paralysis) to 5 (normal) function for each muscle. Because 10 muscles are being tested (5 in each leg), the total possible motor score is 50.
  units on a scale | 34.2 (11.5) | 36.2 (8.4) | 34.8 (10.3)
Body Mass [Mean (Standard Deviation); unit: kg] — Body mass was determined from a DXA (dual energy x-ray absorptiometry) assessment prior to the 3-month intervention.
  kg | 80.8 (14.6) | 94.3 (25.0) | 85.3 (19.1)
ASIA Impairment Scale [Number; unit: participants] — American Spinal Injury Association (ASIA) Impairment Scale is used to grade the degree of sensory & motor impairment.
  ASIA impairment scale C- motor function preserved below the neurological level with > half of the key muscles below the neurological level displaying a grade of less than 3 on a 5-pt scale.
  ASIA impairment scale D- motor function is preserved below the neurological level with at least half of the key muscles below the neurological level displaying a grade of 3 or more on the 5-pt scale.
  for neurological level see: http://asia-spinalinjury.org/elearning/ASIA_ISCOS_high.pdf
  participants
    ASIA impairment C | 2 | 0 | 2
    ASIA impairment D | 10 | 6 | 16
Impairment Function [Number; unit: participants] — Tetraplegia- refers to impairment or loss of function in the cervical region with an effect to the upper and lower extremity
  Paraplegia- impairment or loss of function to the thoracic, lumbar, or sacral regions with an effect to the lower extremity
  participants
    Tetraplegia | 8 | 6 | 14
    Paraplegia | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Cardiovascular Fitness as Determined by Lokomat Peak VO2 Assessments
Description: Peak V02 measurements taken during Lokomat exercise in order to measure cardiovascular fitness.
  Please note that at times the home stretching group would have a second set of measurements at 3 months - one post the 3 month time interval and one later in the 3rd month if there was some delay in initiating the crossover to Lokomat training. This sometimes occurred if the time it would take to complete all of the required studies (e.g. DXA, other secondary measures) was prolonged because of logistical issues.
Time Frame: 0, 1.5 and 3, 4.5, and 6 months
Population: A single outlier point in the baseline data in one control subject was noted. Laboratory journal notes for this subject indicated that this individual had far more episodes of robotic treadmill stops during his baseline testing due to a high degree of spasticity. Given this, we felt justified in excluding this outlier from further data analysis.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Home Stretching Then Lokomat Training: Patients will participate in a home stretching program for 3 months.
  Home stretching protocol : Patients will be instructed by a physical therapist on how to perform a home stretching protocol 3 times per week for 3 months. The stretching will be monitored via telephone by the study coordinator. This will be an active control arm.
  The stretching group will cross-over to the exercise intervention after completion of the 3-month home-base phase. At that time, they will receive an exercise treatment in the Lokomat device 3 times per week for 3 months. Each session will last approximately 45 minutes.
Arm/Group | Lokomat Training | Home Stretching Then Lokomat Training
Number analyzed (Participants) | 12 | 6
ml/kg/min
  Pre (time frame 0) VO2 peak | 20.2 (7.4) | 12.9 (4.4)
  Midpoint (1.5 months) VO2 peak | 22.5 (7.9) | 11.6 (5.1)
  Post_VO2 peak (3 months) | 22.7 (7.5) | 13.4 (3.9)
  Home stretch group at 3 months pre Lokomat (n=6) | NA (NA) — Treatment completed | 18.7 (8.6)
  Home stretch group VO2 peak midpoint (4.5 months) | NA (NA) — Treatment completed | 19.3 (8.4)
  Home stretch group VO2 peak post (6 months) | NA (NA) — Treatment completed | 18.7 (7.0)

2. Secondary Outcome: Body Mass
Description: DXA assessment of total body mass.
  Please note that at times the home stretching group would have a second set of measurements at 3 months - one post the 3 month time interval and one later in the 3rd month if there was some delay in initiating the crossover to Lokomat training. This sometimes occurred if the time it would take to complete all of the required studies (e.g. DXA, other secondary measures) was prolonged because of logistical issues.
Time Frame: Measured at Baseline (Time point 0), 3, and 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lokomat Training | Home Stretching Then Lokomat Training
Number analyzed (Participants) | 12 | 6
kg
  Body Mass_Baseline | 80.8 (14.6) | 94.3 (25.0)
  Body Mass_Post (3 months) | 79.8 (15.0) | 92.3 (23.3)
  Home stretch group pre (3 months) Body mass | NA (NA) — Treatment completed | 93.4 (22.8)
  Home stretch group post Body mass (6 months) | NA (NA) — Treatment completed | 94.8 (22.1)

3. Secondary Outcome: Percent Body Fat
Description: An assessment of percent body fat as determined by DXA analysis.
  Please note that at times the home stretching group would have a second set of measurements at 3 months - one post the 3 month time interval and one later in the 3rd month if there was some delay in initiating the crossover to Lokomat training. This sometimes occurred if the time it would take to complete all of the required studies (e.g. DXA, other secondary measures) was prolonged because of logistical issues.
Time Frame: Measured at Baseline (Time point 0), 3, and 6 months
Measure: Mean (Standard Deviation); unit: percent of total mass
Arm/Group | Lokomat Training | Home Stretching Then Lokomat Training
Number analyzed (Participants) | 12 | 6
percent of total mass
  Percent Body Fat_Baseline (time 0) | 33.6 (7.9) | 34.2 (6.9)
  Percent Body Fat_Post (3 months) | 32.4 (7.7) | 33.3 (7.4)
  Home stretch group pre %Body fat (3 months) | NA (NA) — Treatment completed | 33.3 (7.2)
  Home stretch group post %Body fat (6 months) | NA (NA) — Treatment completed | 33.7 (6.4)

4. Primary Outcome: Cardiovascular Fitness as Determined by Arm Cycle Ergometry VO2 Peak Assessments.
Description: Peak oxygen consumption during arm cycle ergometry as a measure of cardiovascular fitness.
  Please note that at times the home stretching group would have a second set of measurements at 3 months - one post the 3 month time interval and one later in the 3rd month if there was some delay in initiating the crossover to Lokomat training. This sometimes occurred if the time it would take to complete all of the required studies (e.g. DXA, other secondary measures) was prolonged because of logistical issues.
Time Frame: 0, 1.5 and 3, 4.5, and 6 months
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Lokomat Treatment: Subjects will receive active exercise treatment in the Lokomat device 3 times per week for 3 months. Each session will last approximately 45 minutes.
  Lokomat Training : The Lokomat is a robotically assisted partial weight suspension treadmill training device that has the potential to restore leg function in persons with incomplete leg paralysis.
Arm/Group | Lokomat Treatment | Home Stretching Then Lokomat Training
Number analyzed (Participants) | 12 | 6
ml/kg/min
  Pre (time frame 0) VO2 peak arm ergometry | 20.0 (6.5) | 13.5 (3.3)
  Midpoint (1.5 months) VO2 peak arm ergometry | 19.8 (5.4) | 11.1 (2.1)
  Post (3 months) VO2 peak arm ergometry | 21.7 (7.5) | 13.7 (2.5)
  Home stretch group (3 months) pre Lokomat training | NA (NA) — Treatment completed | 13.2 (2.9)
  Home stretch group midpoint (4.5 m) Lokomat | NA (NA) — Treatment completed | 12.3 (5.0)
  Home stretch group post Lokomat (6 mod) | NA (NA) — treatment completed | 13.0 (4.1)

5. Secondary Outcome: Lean Muscle Mass
Description: DXA measurement of total lean muscle mass.
  Please note that at times the home stretching group would have a second set of measurements at 3 months - one post the 3 month time interval and one later in the 3rd month if there was some delay in initiating the crossover to Lokomat training. This sometimes occurred if the time it would take to complete all of the required studies (e.g. DXA, other secondary measures) was prolonged because of logistical issues.
Time Frame: Measured at Baseline (Time point 0) and 3 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lokomat Training | Home Stretching Then Lokomat Training
Number analyzed (Participants) | 12 | 6
kg
  Lean Muscle Mass_Baseline (0 months) | 51.2 (8.5) | 58.9 (11.3)
  Lean Muscle Mass_Post (3 months) | 51.4 (8.0) | 58.3 (9.6)
  Home stretch Group Pre Lean Muscle Mass (3 months) | NA (NA) — Treatment completed | 59.0 (9.5)
  Home muscle Group Post Lean Muscle Mass (6 months) | NA (NA) — Treatment completed | 59.9 (10.2)

6. Secondary Outcome: Bone Mineral Content
Description: DXA assessment of bone mineral content.
  Please note that at times the home stretching group would have a second set of measurements at 3 months - one post the 3 month time interval and one later in the 3rd month if there was some delay in initiating the crossover to Lokomat training. This sometimes occurred if the time it would take to complete all of the required studies (e.g. DXA, other secondary measures) was prolonged because of logistical issues.
Time Frame: Measured at Baseline (Time point 0), 3, and 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lokomat Training | Home Stretching Then Lokomat Training
Number analyzed (Participants) | 12 | 6
kg
  Bone Mineral Content_Baseline (0 months) | 3.04 (0.46) | 3.18 (0.46)
  Bone Mineral Content_Post (3 months) | 3.02 (0.44) | 3.16 (0.55)
  Home stretch Pre Bone Mineral Content (3 months) | NA (NA) — Treatment completed | 3.17 (0.56)
  Home stretch Post Bone Mineral Content (6 months) | NA (NA) — Treatment completed | 3.15 (0.50)

7. Secondary Outcome: Six Minute Walk
Description: A functional capacity test to evaluate walking distance during a 6-minute time frame.
  This measure was only done on those participants that were able to walk for 6 minutes, which represented 9 in the Lokomat training group out of the 12 total randomized to Lokomat training, and 5 out of the 6 randomized to the home stretching group.
  Please note that at times the home stretching group would have a second set of measurements at 3 months - one post the 3 month time interval and one later in the 3rd month if there was some delay in initiating the crossover to Lokomat training. This sometimes occurred if the time it would take to complete all of the required studies (e.g. DXA, other secondary measures) was prolonged because of logistical issues.
Time Frame: Measured Baseline (Time point 0) and 3 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Lokomat Training | Home Stretching Then Lokomat Training
Number analyzed (Participants) | 9 | 5
meters
  Six-minute Walk_Baseline (0 months) | 179.5 (76.4) | 203.0 (108.3)
  Six-minute Walk_Post (3 months) | 201.6 (94.6) | 250.8 (136.3)

8. Secondary Outcome: 10-meter Walk
Description: A functional capacity test to measure speed.
  This measure was only done on those participants that were able to walk, which represented 9 in the Lokomat training group out of the 12 total randomized to Lokomat training, and 5 out of the 6 who were randomized to home stretching.
  Note that at times the home stretching group would have a second set of measurements at 3 months - one post the 3 month time interval and one later in the 3rd month if there was some delay in initiating the crossover to Lokomat training. This sometimes occurred if the time it would take to complete all of the required studies (e.g. DXA, other secondary measures) was prolonged because of logistical issues.
Time Frame: Measured at Baseline (Time point 0) and 3 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Lokomat Training | Home Stretching Then Lokomat Training
Number analyzed (Participants) | 9 | 5
seconds
  10-meter walk_Baseline (0 months) | 23.0 (17.5) | 16.5 (7.6)
  10-meter walk_post (3 months) | 21.3 (17.8) | 14.6 (7.1)

9. Secondary Outcome: Step Activity Monitor
Description: The step activity monitor measures the total steps taken by an individual over a 48 hour time frame in the home environment.
  This measure was only done on those participants that were able to walk in the community and did not use a wheelchair for community mobility, which represented 7 in the Lokomat training group out of the 12 total randomized to Lokomat training and 5 out of 6 of the people randomized to home stretching.
  Please note that at times the home stretching group would have a second set of measurements at 3 months - one post the 3 month time interval and one later in the 3rd month if there was some delay in initiating the crossover to Lokomat training. This sometimes occurred if the time it would take to complete all of the required studies (e.g. DXA, other secondary measures) was prolonged because of logistical issues.
Time Frame: Measured at Baseline (Time point 0) and 3 months
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Lokomat Training | Home Stretching Then Lokomat Training
Number analyzed (Participants) | 7 | 5
steps
  Average 24-hour step total_Baseline (0 months) | 1674.8 (1129.1) | 1531.3 (1576.2)
  Average 24-hour step total_Post (3 months) | 1579.9 (1078.4) | 1652.4 (1707.1)

ADVERSE EVENTS:
Groups:
- Home Stretching Then Lokomat Training: Patients will participate in a home stretching program for 3 months.
  Home stretching protocol : Patients will be instructed by a physical therapist on how to perform a home stretching protocol 3 times per week for 3 months. The stretching will be monitored via telephone by the study coordinator. This will be an active control arm.This group will switch to the 3-month robotic intervention after completing the home-based training program.
Arm/Group | Lokomat Training | Home Stretching Then Lokomat Training
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/6
Other Adverse Events (participants affected / at risk) | 5/15 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lokomat Training (N=15) | Home Stretching Then Lokomat Training (N=6)
Chest and Abdominal Pain (Cardiac disorders) | 1 (1) | 0 (0) — EKG was not consistent with cardiac ischemia. The subject was excluded from further exercise until he was able to undergo a thallium stress test, which did not reveal any ischemic cardiovascular disease
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lokomat Training (N=15) | Home Stretching Then Lokomat Training (N=6)
Skin abrasion (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) — Participants experienced skin abrasions in several areas due to the parachute harness. The following areas were affected: scrotum, scapulae, leg, axilla, chest, shoulder, and groin
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 0 (0) | 1 (2) — One participant experienced several urinary tract infections during the course of the study.
Bruise (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) — The participant experienced a bruise to the sternum and groin regions on 2 separate visits
General pain and lethargy (General disorders) | 1 (1) | 1 (1) — Several participants experienced general skeletal muscle, back and knee pain
Blood in urine (Renal and urinary disorders) | 1 (1) | 0 (0) — The participant observed blood in his urine. The participant was referred to his urologist for evaluation. This incident did not affect the participant's involvement in the training intervention.
Hypotensive response (General disorders) | 1 (1) | 0 (0) — The participant began to experience dizziness and light-headed symptoms prior to a training intervention. A low blood pressure response may have been factor for this event
Significant Weight Loss (General disorders) | 0 (0) | 1 (1) — The participant reported a 20 pound with loss during a 3-4 month time frame. The participant was instructed to schedule an appointment with his primary care physician for a complete evaluation.
Ankle Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The participant reported ankle swelling following a 45-minute robotic training session. The research medical staff evaluated the problem and cleared the participant to continue training with minimal limitations to the exercise intensity and duration.

LIMITATIONS AND CAVEATS:
1. Skin irritation caused missed sessions.
2. Attendance rates were lower than desired given medical and transportation factors.
3. No clearly defined exclusion criteria for bone density in individuals with SCI using this type intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No